CLINICAL TRIAL: NCT05836493
Title: Very Long-term (>15 Years) Results of Tricuspid Valve Repair.
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: VLT-TVR
Record Dates: First submitted 2023-01-27; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ring annuloplasty
  Interventions: Procedure: Ring annuloplasty
- Suture procedure
  Interventions: Procedure: Suture procedure

INTERVENTIONS:
Procedure: Ring annuloplasty — A prosthetic ring is implanted to treat tricuspid regurgitation
  Groups: Ring annuloplasty
Procedure: Suture procedure — Suture techniques such as Kay or De Vega are used to reduce tricuspid annulus in order to treat tricuspid regurgitation
  Groups: Suture procedure

SUMMARY:
Interest in Tricuspid valve disease grew exponentially in the last years in response to an increased awareness of the poor outcome of patients with functional Tricuspid Regurgitation (TR). Earlier reports advocated for a more conservative TR management in patients undergoing left-sided heart valve surgery but more recent guidelines advised for a more aggressive TR management, as accumulating evidence demonstrates its adverse impact on long term morbidity and mortality. Several papers have been published analyzing the results of surgical tricuspid valve repair but the length of the follow-up is usually limited to 10 to 12 years. With this study the investigators aim to analyze the very long-term results (>15years) of tricuspid valve repair according to the surgical method employed for valve repair (suture vs ring annuloplasty).

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgery treatment of TR, isolated or in conjunction with other procedures on the left heart
* patients operated on between January 1998 and December 2004

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - patients operated for non-valvular procedures (e.g. coronary artery bypass)
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, a minimum of 15 years

SECONDARY OUTCOMES:
Reintervention | through study completion, a minimum of 15 years
TR recurrence | through study completion, a minimum of 15 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No